CLINICAL TRIAL: NCT02684630
Title: A Multicenter Study to Evaluate Modified Postcount Algorithm Software on the Trima Accel® System in Volunteer Blood Donors
Brief Title: Trima Accel® System Post Count Algorithm Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CTS-5054
Record Dates: First submitted 2015-11-03; First posted 2016-02-18 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Platelet Product (Experimental): Healthy adult volunteer blood donors that qualify for a single unit platelet collection, with or without other components, will undergo plateletpheresis on the Trima Accel® Automated Blood Collection System (Trima Accel System).
  Interventions: Device: Trima Accel System
- Double Platelet Product (Experimental): Healthy adult volunteer blood donors that qualify for a double unit platelet collection, with or without other components, will undergo plateletpheresis on the Trima Accel® Automated Blood Collection System (Trima Accel System).
  Interventions: Device: Trima Accel System

INTERVENTIONS:
Device: Trima Accel System — Platelet Apheresis Procedure

SUMMARY:
The purpose of this study is to optimize collected platelet yields in single and double platelet collections, while maintaining donor postplatelet count of >100,000/µL.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-randomized study to evaluate Trima Accel System modified postcount algorithm software.

Platelets will be collected according to the Trima Accel System Operator's Manual. Collection procedures will include those in which:

1. a single platelet product is collected
2. a double platelet product is collected, with or without other components.

Study participation will be up to 8 days. The apheresis procedure can last from 25 to 150 minutes, dependent upon the product(s) to be collected, machine configuration, donor parameters, the quality of the vascular access, and the tolerance of the donor to the citrate anticoagulant.

Donors will have one apheresis procedure and follow-up with any serious adverse events for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Meets Blood Center criteria for blood donation and is scheduled for an apheresis procedure that includes a single or double platelet product. These criteria are based on FDA Regulations and American Association of Blood Banks (AABB) Guidelines.
* Appears to have adequate venous access to obtain a postprocedure platelet count.
* Has given written informed consent.

Exclusion Criteria:

* Has undergone a splenectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01-28; Primary Completion 2016-05-28 (Actual); Study Completion 2016-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Pidcoke, MD, PhD, Study Director — Terumo BCT, Inc
Locations (2):
- United States (2):
  - San Diego Blood Bank, San Diego, California
  - Bonfils Blood Center, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 131 volunteers signed consent and were enrolled, but 3 were screen fails and therefore did not participate in the study
Groups:
- Single Platelet Product: Healthy adult volunteer blood donors that qualify for a single unit platelet collection, with or without other components, will undergo plateletpheresis on the Trima Accel System.
  Trima Accel System: Platelet Apheresis Procedure
- Double Platelet Product: Healthy adult volunteer blood donors that qualify for a double unit platelet collection, with or without other components, will undergo plateletpheresis on the Trima Accel System.
  Trima Accel System: Platelet Apheresis Procedure
Period: Overall Study
Arm/Group | Single Platelet Product | Double Platelet Product
Started | 65 | 63
Completed | 60 | 60
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: The Safety Population was used to evaluate participant demographics and treatment emergent adverse events (TEAE).
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Platelet Product | Double Platelet Product | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Customized [Count of Participants; unit: Participants]
  Age ≥ 18 years | 65 | 63 | 128
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 42 | 46 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  Black | 2 | 2 | 4
  Hispanic | 3 | 5 | 8
  White | 56 | 53 | 109
  Other | 1 | 1 | 2
  Unknown | 2 | 0 | 2
Height (in) [Mean (Standard Deviation); unit: inches] | 68.9 (3.95) | 69.0 (3.43) | 69.0 (3.69)
Weight (lbs) [Mean (Standard Deviation); unit: pounds] | 190.3 (37.59) | 191.6 (31.23) | 191.0 (34.47)
Total Blood Volume (mL) [Mean (Standard Deviation); unit: mililiters] | 5214.3 (905.93) | 5285.7 (735.86) | 5249.5 (824.15)

OUTCOME MEASURES:

1. Primary Outcome: Donor Postprocedure Platelet Count Following Donation of Single Platelet Product
Description: The primary endpoint for this study was the postprocedure participant platelet count for participants who have completed a single or double platelet collection. A procedure was a success if the participant's postprocedure platelet count was ≥ 100,000 platelets/μL. A procedure was a failure if the participant's postprocedure platelet count was < 100,000 platelets/μL.
Time Frame: The blood draw to determine postprocedure platelet count will occur ≥ 15 minutes after the end of apheresis
Population: The Full Analysis Set (FAS) included all participants that completed the study and did not meet any of the protocol exclusion criteria. A participant could only have 1 product included in the FAS. The FAS was used to examine the primary and secondary endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Platelet Product | Double Platelet Product
Number analyzed (Participants) | 60 | 60
Participants
  Success (n) | 60 | 60
  Failure (n) | 0 | 0
Statistical Analysis 1: Comparison: Single Platelet Product; Sample Size Determination: Up to 160 participants were to be enrolled in this study to ensure 60 evaluable single platelet product collections and 60 evaluable double platelet product collections. This number was chosen to meet the FDA requirements of 95% of postprocedure participant platelet count of ≥ 100,000 platelets/μL with 95% confidence; Test type: Other — A procedure is a success if the donor's post-procedure platelet count is ≥ 100,000 platelets/μL, lower one-sided 95% confidence interval for the procedure success rate is at least 95%; Simple sample proportion = 1.00, 95% CI 1-sided [lower limit 0.951], Standard Deviation 0 — Estimated proportion is 100%. Hence standard deviation is estimated as 0

2. Primary Outcome: Donor Postprocedure Platelet Count Following Donation of Double Platelet Product
Description: The primary endpoint for this study was the participant's postprocedure platelet count after completing a double platelet collection. A procedure was considered a success if the participant's postprocedure platelet count was ≥ 100,000 platelets/μL.
Time Frame: The blood draw to determine post procedure platelet count will occur ≥ 15 minutes after the end of apheresis
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Single Platelet Product | Double Platelet Product
Number analyzed (Participants) | 60 | 60
Participants
  Success (n) | 60 | 60
  Failure (n) | 0 | 0
Statistical Analysis 1: Comparison: Double Platelet Product; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Simple sample proportion = 1.00, 95% CI 1-sided [lower limit 0.951], Standard Deviation 0 — Estimated proportion is 100%. Hence standard deviation is estimated as 0

ADVERSE EVENTS:
Time Frame: Adverse events that occurred during and up to 24 hours after the apheresis procedure were recorded.
Arm/Group | Single Platelet Product | Double Platelet Product
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/63
Other Adverse Events (participants affected / at risk) | 5/65 | 2/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Platelet Product (N=65) | Double Platelet Product (N=63)
Citrate Toxicity (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Metabolism and nutrition disorders including overall and citrate toxicity.
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) — Nervous system disorders including paraesthesia.
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) — Nervous system disorders including presyncope.
Injection Site Extravasation (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions including injection site extravasation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No